CLINICAL TRIAL: NCT03862287
Title: Is Lidocaine Really Guilty? A Prospective, Randomized, Double Blind Comparison of the Incidence of TNS After Intrathecal Lidocaine Administration vs. Intrathecal Bupivacaine in Patients Undergoing Spinal Anesthesia
Brief Title: Incidence of TNS After Intrathecal Lidocaine v.s Bupivacaine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, JF Asenjo, Professor of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-4823
Record Dates: First submitted 2019-02-19; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Orthopedic Disorder; Leg Injuries
MeSH Terms: conditions — Musculoskeletal Diseases; Leg Injuries | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Lidocaine (Active Comparator): Patients will receive spinal anesthesia in the sitting position under strict sterile conditions in the operating room. Using a median or paramedian approach, the spinal needle will be inserted into the L2-3 or L3-4 interspace to reach the subarachnoid space. After confirming the space by free flow of CSF, 60 mg of isobaric preservative-free Lidocaine 2% will be injected. Sedation using propofol infusion (50-100 mcg/kg/min) and fentanyl (0.5-1 mcg/kg) will be given throughout the procedure as required.
  Interventions: Drug: Lidocaine
- Intrathecal Bupivacaine (Active Comparator): Patients will receive spinal anesthesia in the sitting position under strict sterile conditions in the operating room. Using a median/paramedian approach, the spinal needle will be inserted into the L2-3 or L3-4 interspace to reach the subarachnoid space. After confirming the space by free flow of CSF, 6 mg of 0.5% isobaric bupivacaine will be injected. Sedation using propofol infusion (50-100 mcg/kg/min) and fentanyl (0.5-1 mcg/kg) will be given throughout the procedure as required.
  Interventions: Drug: Bupivacaine Hcl 0.5% Inj_#2

INTERVENTIONS:
Drug: Lidocaine — See arm description.
  Arms: Intrathecal Lidocaine
Drug: Bupivacaine Hcl 0.5% Inj_#2 — See arm description.
  Arms: Intrathecal Bupivacaine

SUMMARY:
This study will look into the incidence of Transient neurological symptoms (TNS) after the intrathecal use of lidocaine in comparison to intrathecal Bupivacaine.

DETAILED DESCRIPTION:
Ever since the introduction of Spinal anesthesia in 1898 by the German surgeon August Bier, the approach gained wide acceptance by the anesthesia community 1. Since that time, the technique has evolved to accommodate a wide variety of surgical procedures, making it one of the most common regional anesthesia modalities used. The advancement of the anesthesia field has led to the advancement of the technique it self, specially the drugs used in it.

A wide range of local anesthetics has been introduced after the initial successful intrathecal use of cocaine. Starting with amylocaine, and later with the introduction of various local anesthetics such as procaine, 2-chloroprocaine, lidocaine, tetracaine, mepivacaine, prilocaine, bupivacaine, with ropivacaine and levobupivacaine being introduced last. Many of these drugs have fallen out of favour due to various reasons, with Lidocaine, procaine, mepivacaine, ropivacaine and bupivacaine still being used in clinical practice 2.

The choice of the local anesthetic used depends on many factors such as the duration of the operation, the type of surgery and the degree of motor blockade desired. With the advancement of surgery and the increase in day surgical cases, a need for a fast acting, short in duration local anesthetic that allows fast recovery and early discharge has emerged. Of all the local anesthetic drugs available, Lidocaine is one of the drugs that fulfills these needs.

Common complications associated with the use of this technique include headache (5%), backache (11%), hypotension, bradycardia, nausea and vomiting (20%), urinary retention, hypothermia and transient neurological syndrome (TNS). More serious complications include total spinal, infection (meningitis/ encephalitis) and epidural hematoma (<1 in 150,000). On the other hand, complications related to receiving General Anesthesia for the same procedure are similar, with higher chances of nausea and vomiting or airway problems.

TNS is defined as back pain and/or dysesthesia radiating bilaterally to the legs or buttocks after total recovery from spinal anesthesia, manifesting within 24 hours after the surgery and typically lasting less than a week. The etiology of TNS is unknown. Possible contributing factors to the development of TNS include sciatic nerve stretching causing neural ischemia, vasoconstriction of spinal cord arteries, patient positioning, direct needle injury and pooling of local anesthetic in the sacral region. The pathophysiology of TNS is unknown, and there is no specific lab test to diagnose this complication. Treatment of TNS, includes bed rest, administration of nonsteroidal anti inflammatory drugs and sometimes the addition of an opioid is needed 3.

All local anesthetics have been shown to cause TNS, with lidocaine appearing to have the greatest risk. The first reported case of TNS after the single shot administration of 5% hyperbaric lidocaine was published by Schneider and colleagues in 1993 4, which was confirmed later by several other studies 5-9. The reported incidence of TNS after the administration of lidocaine ranges from 10%-40% 10-13. In a more resent study done by F. Salazar et al. the incidence of TNS with lidocaine was reported to be 2.5%, much lower than what was previously described in the literature 14.

Furthermore, in an internal audit done at the MGH looking at all spinal anesthesia cases performed by Dr. Asenjo in the past two years, TNS incidence was found to be 2.7%, far less than what the literature describes, and correlates more with what F. Salazar et al. found in their study. We want to clarify this discrepancy in the incidence of TNS with lidocaine since this is a very inexpensive agent, with a short to intermediate duration of action and readily available world wide. With this purpose we have designed a randomized controlled trial to test the hypothesis that the incidence of TNS after spinal anesthesia with lidocaine is much lower than what was previously described in the literature. This trial will also look at the natural course of the symptoms of TNS.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III male and female patients aged between 18 to 80 years old, who will receive spinal anesthesia for surgeries lasting less than one hour.

Exclusion Criteria:

* Patients younger than 18 years old.
* ASA physical status >3.
* Immunosuppression or high risk of infection.
* Contraindications to receiving spinal anesthesia (e.g. coagulation impairment).
* Patients with psychosis
* Patients with preexisting back pain.
* Patients with cognitive impairment
* Allergies to local anesthetics, analgesics or any medication used in the study.
* Patients with chronic regular opioid usage
* Presence of preexisting neurological symptoms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Transient Neurological Symptoms | Day 1
  To determine the incidence of TNS following the use of intrathecal Lidocaine as compared with Bupivacaine
Transient Neurological Symptoms | Day 3
  To determine the incidence of TNS following the use of intrathecal Lidocaine as compared with Bupivacaine

SECONDARY OUTCOMES:
Transient Neurological Symptoms | Day 1 and day 3 postoperative
  To determine the incidence of TNS following the use of intrathecal Bupivacaine
Transient Neurological Symptoms | Day 1 and day 3 postoperative
  To determine the incidence of TNS following the use of either intrathecal Lidocaine and Bupivacaine in patients operated in the lithotomy position

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF